CLINICAL TRIAL: NCT02440971
Title: Adaptive Servo Ventilation (ASV) in the Management of Acute Decompensated Heart Failure (ADHF)
Brief Title: Adaptive Servo Ventilation (ASV) in Heart Failure
Status: Suspended | Type: Observational
Sponsor: St Vincent's University Hospital, Ireland (Other)
Collaborators: ResMed (Industry)
Responsible Party: Principal Investigator, Mark Ledwidge, Professor Ken McDonald, Consultant Cardiologist, St Vincent's University Hospital, Ireland, St Vincent's University Hospital, Ireland
Other Study IDs: HFU-CM-001
Record Dates: First submitted 2013-12-23; First posted 2015-05-12 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Acute Decompensated Heart Failure; Sleep Disordered Breathing
Keywords: Adaptive Servo Ventilation; Acute decompensated heart failure; SleepMinder; ApneaLink Plus; Sleep disordered breathing; Natriuretic peptide
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: S9-Autoset CS-A — The S9-Autoset CS-A is an adaptive servo-ventilation (ASV) machine. It adjusts the level of inspiratory support automatically in response to the patient's respiratory effort. Inspiratory support is increased in the presence of hypoventilation and decreased in the presence of hyperventilation.

SUMMARY:
Up to 60% of patients with heart failure show abnormal patterns of breathing (sleep disordered breathing (SDB)) at night which can increase the risk of recurrent admissions and have important prognostic implications. SDB is however, treatable with the use of non invasive breathing support devices such as the adaptive servo ventilation (ASV) device. The aim of the study is to observe and investigate the potential role of ASV in the management of heart failure.

Patients that agree to participate in this study will be requested to use an ASV ventilator device (called the AutoSet CS-A) to help their SDB for approximately 6 weeks. The device is approximately the size of a large shoe box, which can be placed at the side of the bed, with tubing and a mask. At night, the mask is placed over the nose and/or mouth and it blows positive air pressure as determined by the device itself as it constantly monitors the patients breathing throughout the night. During this study, the patients breathing patterns will be monitored non-invasively using the ApneaLink device. A non-contact device knows as a SleepMinder will sit on the patients bedside locker as another form of monitoring of their sleep patterns. Study staff will monitor the patient and give them frequent support, and they will also be asked questions regarding their experiences with this equipment and any symptoms they may have over this time. They will be followed up regarding this study at the same time as their follow-up requirements for their heart failure. This study will be conducted in total over 3 months.

DETAILED DESCRIPTION:
Sleep disordered breathing (SDB) is common in patients with heart failure (HF) and is an independent predictor of morbidity and mortality. Adaptive servo-ventilation (ASV) is reported as the most effective treatment for SDB in HF and has been shown to improve cardiac function in patients with HF coexistent with SDB. ASV may also be an effective therapeutic option for patients with HF regardless of presence or severity of SDB.

The aim of the study is to investigate the potential role for ASV in improving the management of ADHF in the acute hospital phase and reducing complications in the vulnerable post discharge period. This is an observational study of forty patients admitted to hospital with ADHF.

In this clinical investigation, the ApneaLinkTM Plus device will measure patient respiratory nasal airflow, snoring, blood oxygen saturation, pulse and respiratory effort during sleep. The research participant will be connected to the device during their inpatient hospitalisation as soon as they are stabilised off oxygen. These recordings will aid the diagnosis of SDB for further clinical investigation.

The S9 Autoset CS-A system will be evaluated to determine whether ASV has beneficial effects on the cardiac function of patients with ADHF. During an in-patient run-in phase, the patients tolerability to ASV therapy will be assessed and if tolerated well, the patient will continue with this therapy following discharge for 45 days.

The SleepMinder sensor device will monitor the sleep and breathing patterns of the participants as they sleep, and in doing so, sleep apnoeas will be detected. Each patient will monitor their weight daily using a Precision Personal Health Scales for 90 days. Finally, a questionnaire will be completed by the patient which allows them to self-report their HF symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the hospital with a primary diagnosis of ADHF
* Stable off oxygen for 24 hours
* Informed consent
* Age ≥ 18 years

Exclusion Criteria:

* Age < 18 years
* Pregnant women, breastfeeding mothers
* Anyone not capable of giving informed consent
* Contraindications to positive airway pressure:

  * Severe bullous lung disease
  * Dehydration
  * Cerebrospinal fluid leak
  * Acute sinusitis or otitis media
  * Epistaxis (severe nose bleeds) causing a risk of pulmonary aspiration
  * Conditions predisposing to a risk of vomiting into mask
  * Impaired ability to clear secretions
  * Hypotension (defined as systolic BP < 100mmHg) or significant intravascular volume depletion
  * Pneumothorax or pneumomediastinum
  * Recent cranial trauma or surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted into hospital for acute management of ADHF are eligible to participate in this study (providing inclusion/exclusion criteria are met)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-05; Primary Completion 2019-05 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Length of inpatient HF hospitalisation | Patients are followed during the inpatient admission, currently an average of 14 days
  Admission to ready-for-discharge in days
Time to clinical stability (days) | Patients are followed during the inpatient admission and an approximate time to clinical stability is determined, currently less than an average of 14 days

SECONDARY OUTCOMES:
Time to event using a combined morbidity index | From baseline to study end, an average of approximately 12 months
  Time to event using a combined morbidity index including re-hospitalisation (all-cause, cardiac, HF), outpatient attendance with intravenous diuretics, outpatient attendance with symptomatic deteriorations requiring adjustment of oral diuretic, home/patient adjustment of oral diuretic treatment without patient outpatient clinic attendance.
Natriuretic peptide (NTproBNP) levels | Baseline, 45 days and 90 days
B-Type Natriuretic peptide (BNP) levels | Baseline, 45 days and 90 days
Ejection fraction | Baseline, 45 days and 90 days
Creatinine clearance | Baseline, 45 days and 90 days
Markers of renal damage | Baseline, 45 days and 90 days
  Kidney injury molecule-1(KIM-1)
Markers of renal damage | Baseline, 45 days and 90 days
  Neutrophil gelatinase-associated lipocalin (NGAL)
Markers of matrix turnover | Baseline, 45 days and 90 days
  Matrix metalloproteinase (MMP)-2 and -9
Markers of inflammation | Baseline, 45 days and 90 days
  hsCRP
Comparative Sleep Disordered Breathing | Baseline, 45 days, 90 days and study end, an average of approximately 12 months
  Measured by the ApneaLinkTM Plus
Comparative Sleep Disordered Breathing | Baseline, 45 days, 90 days and study end, an average of approximately 12 months
  Measured by SleepMinder

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M McDonald, MD, Principal Investigator — St Vincent's University Hospital, Ireland
Locations (1):
- St Vincents University Hospital, Dublin, Ireland